CLINICAL TRIAL: NCT03445663
Title: A Phase 1, First-in-Human, Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 424 in Subjects With Multiple Myeloma
Brief Title: Study Evaluating AMG 424 in Subjects With Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Previous sponsor business decision not to proceed with the AMG 424 asset.
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160445
Record Dates: First submitted 2018-02-01; First posted 2018-02-26 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Relapsed/ Refractory Multiple Myeloma
Keywords: Relapsed/ Refractory Multiple Myeloma; Multiple Myeloma; Oncology/Hematology; Immunotherapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG 424 (Experimental): Comparison of different dosages of AMG 424
  Interventions: Drug: AMG 424

INTERVENTIONS:
Drug: AMG 424 — Subjects will receive IV infusions of AMG 424

SUMMARY:
A multi-center Phase 1, First-in-Human study conducted in 2 Parts, testing AMG 424 in subjects with relapsed/ refractory multiple myeloma.

DETAILED DESCRIPTION:
Part 1 of the study is dose evaluating and aimed at assessing the safety and tolerability of AMG 424 while determining the maximum tolerated dose (MTD) and/or biologically active dose in subjects with relapsed/ refractory multiple myeloma.

Part 2 of the study will further evaluate safety and tolerability of the AMG 424 MTD dose determined in Part 1, in groups of subjects with relapsed/ refractory multiple myeloma that include those with high or low cytogenetic risk.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma meeting the following criteria:
* Pathologically-documented diagnosis of multiple myeloma that has relapsed after at least two prior lines of therapy that must include a proteasome inhibitor (PI), immunomodulatory drug (IMiD), and, where approved and available, anti-CD38 therapy in any order OR that is refractory to PI, IMiD, and anti-CD38 therapy.

  ◾Subjects who could not tolerate a PI, IMiDs, or a CD38-directed therapeutic antibody due to unacceptable toxicities are eligible to enroll in the study.
* Measurable disease as per IMWG response criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2

Exclusion Criteria:

* Known central nervous system involvement by multiple myeloma
* Previously received allogeneic stem cell transplant and one or more of the following:

  * received the transplant < 6 months prior to study Day 1
  * received immunosuppressive therapy < 3 months prior to study Day 1
  * any active acute graft versus host disease (GvHD), grade 2- 4, according to the Glucksberg criteria or active chronic GvHD requiring systemic treatment
  * any systemic therapy against GvHD < 2 weeks prior to study Day 1
* Autologous stem cell transplantation less than 90 days prior to study day 1
* Multiple myeloma with IgM subtype
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Evidence of primary or secondary plasma cell leukemia at the time of screening
* Waldenstrom's macroglobulinemia
* Amyloidosis
* Dexamethasone at cumulative doses of greater than 160 mg or equivalent <3 weeks prior to study Day 1 is not allowed. Use of topical or inhaled steroids is acceptable
* Anticancer treatment (chemotherapy, IMiD, PI, molecular targeted therapy) < 2 weeks prior to study Day 1
* Treatment with a therapeutic antibody targeting CD38 < 12 weeks prior to study Day 1
* Systemic radiation therapy or major surgery < 28 days prior to study Day 1 as well as focal radiotherapy < 14 days prior to study Day 1.
* Major surgery within 28 days prior to study Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Subject incidence of treatment emergent and treatment related adverse events as assessed by CTCAE version 4.0 | 12 Months
  Measure of Safety
Subject incidence of dose limiting toxicities (DLTs) | 28 Days
  Measure of Safety

SECONDARY OUTCOMES:
Anti-tumor activity | 48 Months
  Efficacy parameter measured by IMWG response criteria
Duration of Response | 48 Months
  Measure of Response
Maximum concentration (Cmax) of AMG 424 | 12 Weeks
  Characterize the pharmacokinetic (PK) profile following treatment with AMG 424
Minimum concentration (Cmin) of AMG 424 | 12 Weeks
  Characterize the pharmacokinetic (PK) profile following treatment with AMG 424
Time of maximum concentration (Tmax) of AMG 424 | 12 Weeks
  Characterize the pharmacokinetic (PK) profile following treatment with AMG 424
Area under the concentration-time curve (AUC) of AMG 424 | 12 Weeks
  Characterize the pharmacokinetic (PK) profile following treatment with AMG 424
Time to progression | 48 Months
  Measure of Response
Progression-Free Survival | 48 Months
  Measure of Response
Overall Survival | 48 Months
  Measure of Response

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (6):
  - Research Site, San Francisco, California
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (2):
  - Research Site, Camperdown, New South Wales
  - Research Site, Fitzroy, Victoria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com